CLINICAL TRIAL: NCT03593642
Title: Bilateral Erector Spinae Plane (ESP) Catheters Versus Single Shot ESP Block for Open Heart Surgery in Infants
Brief Title: ESP Catheter Vs Single Shot ESP for Open Heart Surgery in Infants
Acronym: ESPINFANT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vinmec Healthcare System (Other)
Responsible Party: Principal Investigator, Philippe Macaire, Professor in Anesthesiology and Pain, Vinmec Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: vinmechs
Record Dates: First submitted 2018-06-08; First posted 2018-07-20 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Opioid Use; Pain, Postoperative; Quality of Life
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Randomized controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): Erector spinae bilateral catheters with continuous infusion iso saline during 48h after surgery Day 0 to day 2
  Interventions: Drug: Continuous infusion of Iso Saline in ESP catheter
- Regional analgesia group (Experimental): Erector spinae bilateral catheters with continuous infusion Ropivacaine 0.1 or 0.2%, depending on age, infusion during 48h after surgeryDay 0 to day 2
  Interventions: Drug: Continuous infusion of ropivacain in ESP catheter

INTERVENTIONS:
Drug: Continuous infusion of ropivacain in ESP catheter — administration of ropivacaine in ESP catheter to provide regional analgesia after surgery
  Arms: Regional analgesia group
Drug: Continuous infusion of Iso Saline in ESP catheter — administration of Iso Saline in ESP catheter to be the control group
  Arms: Control Group

SUMMARY:
Post operative pain after open heart surgery is still a main concern; current multimodal analgesia modalities have shown good efficacy for postoperative pain at rest, without reaching full pain relief.

The primary goal of this study is to evaluate the effectiveness of peri-operative analgesia, measured by consumption of opioids during the first 48h hours after the surgery, using bilateral erector spinae catheters for 48h, compared to single shot erector spinae block in pediatric patients undergoing open heart surgeries .

DETAILED DESCRIPTION:
Fast track to extubation after pediatric cardiothoracic surgery is becoming more common after a number of reports showing it is safe and effective . However, it has introduced new challenges to pain control. Intubated patients require larger doses of opioids and benzodiazepines for comfort . In patients who are awake and spontaneously breathing, pain and agitation cannot be treated with lower doses.

Some centers still administer continuous infusions of opioid and benzodiazepines to extubated patients. These infusions may not be necessary and may even be harmful.

In a pilot study of adult patients undergoing open heart surgery at VinMec hospitals, peri-operative regional analgesia by continuous bilateral erector spinae plane (ESP) block, Investigators showed that the pain relief was efficient and the requirement for opioids in the first 48 hours post-surgery was zero .

It confirmed that the impact of regional anesthesia techniques on main procedure-specific postoperative outcomes is very important in decreasing opioid use in the context of fast-track recovery programs that are recommended after cardiac surgery.

Since April 2017 Investigators are performing bilateral ESP single shot block in cardiac surgery on infants and children. In the post-operative period the patients still need 30 hours after end of surgery small doses opioids to release their pain according to the evaluation by Comfort-B or/and FLACC Scales after the single shot blocks recovered. Since December 2017 Investigators are performing these surgeries with bilateral ESP catheters with an Intermittent infusion of very low doses of local anesthetic according to the guidelines ] in regional anesthesia analgesia in pediatric to improve the post-operative analgesia and avoid any opioids.

The ESP block is an inter-fascial block described as a quite simple technique, far from risky anatomical structures. Since the first publication in November 2016 only one study on children has been published , in thoracic surgery.

This technique has been presented at the 2018 World Congress on Regional Anesthesia and Pain Medicine as a opioid free pain free for open heart surgery in adult.

Researchers from Stanford University reported also one case in open heart surgery announcing a new era in cardiac anesthesia in adult. A study in press shows the interest of a similar thoracic block named Serratus plane block in thoracic aortic surgery in newborn and infants .

The study will be a double-blind randomized controlled trial. After informed consent from guardians or parents, infants and children will be randomized via a random number generator into one of two treatment groups.

* Group 1 (control) will receive a single shot dose of local anesthestic ropivacaine through ESP catheters and 6 hours later continuous infusion of Iso saline with a rescue analgesia in case of pain.
* Group 2 (treatment) will received a single shot dose of local anesthestic ropivacaine through ESP catheters and 6 hours later a continuous infusion of ropivacaine with a rescue analgesia in case of pain.

Catheter Performance The anesthesia team will check that the catheter is inserted in the inter-fascial space rather than intra-vascular. This procedure will be bilateral. The catheter will have a yellow label on the Huer®-Lock connector to identify clearly that it is regional analgesia catheter to prevent any errors of miss injection. (Yellow is the international identification of regional anesthesia/analgesia lines).

After this control an induction dose is injected according to the pediatric regional anesthesia analgesia guidelines.

* If < 1 year old Ropivacaine 0.1% 0.25 mg/kg/side
* If >= 1 year old Ropivacaine 0.2% 0.50 mg/kg/side

After 7h the ESP catheter has been placed, one of the clinical research nurses will proceed to the randomization of the patient according to the randomization table, and prepare the solution (100 mL) in the pump as per protocol. They will put the ID number of patient on the pump. The nurse will receive instruction to keep strictly confidential the content of the pumps. They will deliver the prepared pumps to the anesthesiologist and anesthesia nurse in charge of the patient. They will connect the pumps to the patient and start the infusion 8 hours after regional anesthesia induction as per protocol.

* Group 1 (control group) will receive an automatic Iso Saline infusion through the 2 ESP catheters. The infusion regimen will be Intermittent automatic bolus (IAB) every 8 hours of 0.5mL/kg/side. The bolus on the second catheter will be delayed by 2 hours.
* Group 2 (Continuous regional analgesia group) will receive an automatic infusion of Ropivacaine (see above for concentration according to age) through the 2 ESP catheters. The infusion regimen will be IAB every 8 hours 0.5mL/kg-side. The bolus on the second catheter will be delayed by 2 hours to reduce the maximal plasmatic concentration as much as possible.

Both groups will receive paracetamol 15 mg/kg every 6 hr.

For all groups pain will be defined according to COMFORT Scale > 17 or FLACC scale > 3.

Management of the pain

1. If pain appears before next IAB the delay between 2 IAB will be reduced to 6 hr without adding any medication This is a common practice in peripheral nerve management.
2. If the block extension is insufficient (T1 to T9) , IAB will be increased by 0,1 mL/catheter of the solution inside the pump on the side concerned: by increasing the volume by 10% Investigators will increase the extension of the analgesia block. This increase in volume will be limited to one increase.

1+ 2/ If pain still persists after 1 hour the patient will be shifted to rescue analgesia described below (3) .

3/ If non of those (1 or 2) patient will receive rescue analgesia start Ibuprofen 10mg/kg/12 h All participants in the studies were trained to the protocol in January 2018; the research nurses were trained to randomization and data collection.

Pain will be reassessed 1 hour after 3a if the FLACC < 3: continue ESP catheters and paracetamol+ ibuprofen /12h if the FLACC >3 = poor analgesia Investigators will add analgesia by opioids as before this technique and commonly used in open heart surgeries in infants o Morphine 30 mcg/kg/h.

A Bi Daily inspection of the catheters insertion points will be done. If redness around puncture point the catheters will be removed and shift to classical IV analgesia to prevent any infection. It will be declared as a minor incident in the study.

ESP catheters will be removed 2 hours after drain removal maximum 46h after insertion.

2 h. after Drain removal and ESP catheter removed the analgesia in both group will be with the following antalgics: Efferalgan : 15-20 mg/kg /6h and Ibuprofen sirop : 10 mg/kg/12h

Pain scales Investigators will use to evaluate the pain:

When patient will be intubated Investigators will use scale Comfort-B . at rest and after pressure on sternum or drain mobilization (Mob).

After extubation and still drains will remain Investigators will use FLACC scale at rest and at Mob (sitting in bed rotation of the thorax) analysis of the Localization of the pain

* Sternum
* Back pain
* Drains o After drains removal Investigators will use FLACC Scale rest and Mob ( sitting in bed rotation of the thorax) and pain localization

One month after the surgery a pain assessment will be done during the 1st one month follow up with a FLACC scale (rest and Mobilisation) and also analyze if the patient is playing normally according to his parents or guardians

Statistical analysis

Based on our prior institutional unpublished retrospective data of morphine consumption in the first 48H after the surgery (End of surgery to 48h after end of surgery) in patients who received Single shot ESP bl0cks who underwent open heart surgeries (control group) (mean 0.998 mg/kg) with standard deviation 0.323) Treated group = 0 mg/kg Investigators determine that a total of 14 patients per arm will be needed to achieve a difference of 0.4 between the 2 groups with 90% power at alpha =0.05. Investigators will assume up to 10% lost to follow up and 10% of patients would be non-compliant so Investigators will enroll 20 patients in each group.

ELIGIBILITY:
Inclusion Criteria:

* Elective open heart surgery

Exclusion Criteria:

* Consent refusal
* Urgent surgery
* unstable hemodynamic patient after anesthesia induction

Ages: 2 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
morphine consumption | 48 hours after arrival in Intensive care unit
  Total consumption of rescue analgesia by morphine (mcg/kg)

SECONDARY OUTCOMES:
pain after extubation at rest | 2 hours after extubation at day 1
  Flacc Scale to evaluate pain in Infants from 0 no pain to 10 maximal pain
pain after extubation at mobilisation seating in the bed | 2 hours after extubation at day 1
  Flacc Scale to evaluate pain in Infants from 0 no pain to 10 maximal pain
Persistent pain at 1 month | Consultation 1 month after the surgery
  Flacc Scale to evaluate pain in Infants from 0 no pain to 10 maximal pain Mobilisation and rest

CONTACTS AND LOCATIONS:
Locations (1):
- Vinmec Central Park, Ho Chi Minh City, Ho Chi Minh, Vietnam

REFERENCES:
- [Background] Garg R, Rao S, John C, Reddy C, Hegde R, Murthy K, Prakash PV. Extubation in the operating room after cardiac surgery in children: a prospective observational study with multidisciplinary coordinated approach. J Cardiothorac Vasc Anesth. 2014 Jun;28(3):479-87. doi: 10.1053/j.jvca.2014.01.003. Epub 2014 Apr 18. PMID 24746595
- [Background] Heinle JS, Diaz LK, Fox LS. Early extubation after cardiac operations in neonates and young infants. J Thorac Cardiovasc Surg. 1997 Sep;114(3):413-8. doi: 10.1016/S0022-5223(97)70187-9. PMID 9305193
- [Background] Kin N, Weismann C, Srivastava S, Chakravarti S, Bodian C, Hossain S, Krol M, Hollinger I, Nguyen K, Mittnacht AJ. Factors affecting the decision to defer endotracheal extubation after surgery for congenital heart disease: a prospective observational study. Anesth Analg. 2011 Aug;113(2):329-35. doi: 10.1213/ANE.0b013e31821cd236. Epub 2011 Apr 13. PMID 21490084
- [Background] Carli F, Kehlet H, Baldini G, Steel A, McRae K, Slinger P, Hemmerling T, Salinas F, Neal JM. Evidence basis for regional anesthesia in multidisciplinary fast-track surgical care pathways. Reg Anesth Pain Med. 2011 Jan-Feb;36(1):63-72. doi: 10.1097/AAP.0b013e31820307f7. PMID 22002193
- [Background] Munoz F, Cubillos J, Bonilla AJ, Chin KJ. Erector spinae plane block for postoperative analgesia in pediatric oncological thoracic surgery. Can J Anaesth. 2017 Aug;64(8):880-882. doi: 10.1007/s12630-017-0894-0. Epub 2017 Apr 26. No abstract available. PMID 28447318
- [Background] Nga Ho, Binh Nguyen, Tan Nguyen, Viet Vu, Chinh Quach, Vincente Rocques, Philippe Macaire Analgesia opioid free with Bilateral ESP catheters for open heart Surgeries in Adults RAPM 2018 ASRA 277
- [Background] Tsui BCH, Navaratnam M, Boltz G, Maeda K, Caruso TJ. Bilateral automatized intermittent bolus erector spinae plane analgesic blocks for sternotomy in a cardiac patient who underwent cardiopulmonary bypass: A new era of Cardiac Regional Anesthesia. J Clin Anesth. 2018 Aug;48:9-10. doi: 10.1016/j.jclinane.2018.04.005. Epub 2018 May 26. No abstract available. PMID 29684728
- [Background] Biswas A, Luginbuehl I, Szabo E, Caldeira-Kulbakas M, Crawford MW, Everett T. Use of Serratus Plane Block for Repair of Coarctation of Aorta: A Report of 3 Cases. Reg Anesth Pain Med. 2018 Aug;43(6):641-643. doi: 10.1097/AAP.0000000000000801. PMID 29794944
- [Background] Referentiels Societe Francaise d'Anesthesie Reanimation (SFAR) ALR pediatrique 2010 and Association des Anesthesistes reanimateurs Pediatriques Francophones ADARPEF http://sfar.org/anesthesie-loco-regionale-en-pediatrie/
- [Result] Alghamdi AA, Singh SK, Hamilton BC, Yadava M, Holtby H, Van Arsdell GS, Al-Radi OO. Early extubation after pediatric cardiac surgery: systematic review, meta-analysis, and evidence-based recommendations. J Card Surg. 2010 Sep;25(5):586-95. doi: 10.1111/j.1540-8191.2010.01088.x. PMID 20626510
- [Derived] Macaire P, Ho N, Nguyen V, Phan Van H, Dinh Nguyen Thien K, Bringuier S, Capdevila X. Bilateral ultrasound-guided thoracic erector spinae plane blocks using a programmed intermittent bolus improve opioid-sparing postoperative analgesia in pediatric patients after open cardiac surgery: a randomized, double-blind, placebo-controlled trial. Reg Anesth Pain Med. 2020 Oct;45(10):805-812. doi: 10.1136/rapm-2020-101496. Epub 2020 Aug 19. PMID 32817407